CLINICAL TRIAL: NCT00940680
Title: A Phase III, 8-week, Multicenter, Randomized, Double-blind Study to Compare the Efficacy and Safety of Amlodipine 5mg+Losartan 100mg Versus Losartan 100mg in Patients With Essential Hypertension Not Controlled on Losartan Monotherapy
Brief Title: Efficacy/Safety of Amlodipine Plus Losartan Versus Losartan in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Director, Hanmi Pharmaceutical Company Limited
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ALOS-302
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Amlodipine; Losartan; hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- amlodipine/losartan 5/100mg (Experimental)
  Interventions: Drug: Amlodipine plus Losartan
- losartan 100mg (Active Comparator)
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Amlodipine plus Losartan — amlodipine/losartan 5/100mg q.d.
  Other Names: Amosartan
  Arms: amlodipine/losartan 5/100mg
Drug: Losartan — losartan 100mg q.d.
  Arms: losartan 100mg

SUMMARY:
The purpose of this study is to evaluate of efficacy and safety of amlodipine plus losartan and losartan alone in patients with essential hypertension inadequately controlled on losartan monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Essential hypertensive patients whose blood pressure is not controlled before the study (sit DBP≥90 mmHg for drug-treated patient, sit DBP≥95mmHg for drug-naïve patient)
* Non-responder to 4 weeks treatment of losartan 100 mg monotherapy (sit DBP≥90mmHg)

Exclusion Criteria:

* mean sit SBP≥200mmHg or mean sit DBP≥120mmHg at screening
* mean sit SBP≥180 mmHg or mean sit DBP≥120mmHg after 4 weeks of losartan 100mg treatment
* has a history of hypersensitivity to dihydropyridines or angiotensin II receptor blockers
* Secondary hypertensive patient or suspected to be
* Uncontrolled diabetes mellitus patients
* Severe heart disease or severe neurovascular disease
* Known as severe or malignant retinopathy
* Patients showed clinically significant hematological finding, patients with renal diseases (serum creatinine), patients with hepatic disease (ALT or AST)
* History of malignancy tumor
* History of autoimmune disease
* History of alcohol or drug abuse
* Positive to pregnancy test, nursing mother, has an intention on pregnancy
* Considered by investigator as not appropriate to participate in the clinical study with othe reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure | Week 8

SECONDARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure | Week 4
Change from baseline in mean sitting systolic blood pressure | Week 4, 8
Responder rate | Week 4, 8

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yun Cho, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- 9 sites in Korea, Seoul, Daegu, Etc., South Korea

REFERENCES:
- [Derived] Hong BK, Park CG, Kim KS, Yoon MH, Yoon HJ, Yoon JH, Yang JY, Choi YJ, Cho SY. Comparison of the efficacy and safety of fixed-dose amlodipine/losartan and losartan in hypertensive patients inadequately controlled with losartan: a randomized, double-blind, multicenter study. Am J Cardiovasc Drugs. 2012 Jun 1;12(3):189-95. doi: 10.2165/11597410-000000000-00000. PMID 22462558